CLINICAL TRIAL: NCT02698462
Title: Adding Family History of Colorectal Cancer to the FIT-based Screening Program in a Dutch Colorectal Cancer Population Sample
Brief Title: Adding Family History of Colorectal Cancer to the Dutch FIT-based Screening Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Evelien Dekker, MD, PhD (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other)
Responsible Party: Sponsor-Investigator, Prof. Evelien Dekker, MD, PhD, Professor MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 821748-140305-PG; TC 12-05 (Other Grant/Funding Number: Dutch Digestive Foundation)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Neoplasms
Keywords: Advanced neoplasia; Colorectal cancer; Population screening; Family history
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FIT and Questionnaire (Other): Six thousand persons eligible for the national CRC screening program will be selected. They will be selected from four areas that are considered representative of the Netherlands. All invitees receive an invitation to complete a FIT (FOB-Gold) and a validated, online family history questionnaire. Answers from the questionnaire are compared with the Dutch criteria for referral for genetic testing and/or surveillance colonoscopies for persons at a potential familial risk for CRC. Invitees are invited to perform both tests, but if they only perform one this will be assessed. Participants with a positive FIT and/or a positive family history and a diagnosis of familial CRC by a clinical geneticist will be referred for colonoscopy.
  Interventions: Other: Family history questionnaire

INTERVENTIONS:
Other: Family history questionnaire — All invitees receive an invitation to complete a FIT (FOB-Gold) and a validated, online family history questionnaire. Answers from the questionnaire are compared with the Dutch criteria for referral for genetic testing and/or surveillance colonoscopies for persons at a potential familial risk for CRC. Invitees are invited to perform both tests, but if they only perform one this will be assessed. Participants with a positive FIT (cut-off value 275 ng/ml) and/or a positive family history and a diagnosis of familial CRC by a clinical geneticist will be referred for colonoscopy.

SUMMARY:
The aim of this study is to identify more persons with advanced neoplasia in the current national CRC screening, by adding data on family history of CRC (using a validated online questionnaire) to FIT. In addition, the aim is to identify those persons and their family members who should not be participating in a FIT based screening but receive surveillance colonoscopies instead, because of a familial CRC syndrome. It is aimed to increase detection without affecting participation, thereby increasing the yield of screening.

DETAILED DESCRIPTION:
This is a prospective CRC population-based screening trial, using FIT and a family history questionnaire, inviting those with a positive FIT, a familial CRC syndrome, or both for colonoscopy.

All invitees receive an invitation to complete a FIT (FOB-Gold) and a validated, online family history questionnaire. Answers from the questionnaire are compared with the Dutch criteria for referral for genetic testing and/or surveillance colonoscopies for persons at a potential familial risk for CRC. Invitees are invited to perform both tests, but if they only perform one this will be assessed. Participants with a positive FIT (cut-off value 275 ng/ml) and/or a positive family history and a diagnosis of familial CRC by a clinical geneticist will be referred for colonoscopy.

The investigators will compare the diagnostic yield, participation rate, and positive predictive value for two strategies: referral for colonoscopy based on FIT and family history versus referral for colonoscopy based on FIT-only.

The sample size is justified by the anticipated gain in diagnostic yield from combining FIT-only with family history screening. With a sample size of 6.000 persons the investigators expect to detect 130 persons with advanced neoplasia after a positive FIT (21.7 per 1.000 invitees). By adding the family history questionnaire, the investigators anticipate detecting an additional number of 11 persons with advanced neoplasia, resulting in a yield of combined FIT-based and family history screening of 141 persons with advanced neoplasia (23.5 per 1.000 invitees), which is an increase of 1.8 per 1.000 invitees. Using the McNemar test with the significance level set at 5%, there is a power of 91% to show that the gain in diagnostic yield is statistically significant. Previous CRC test screening studies using FIT showed that participation rates are approximately 60% in a first screening round. The participation rate in the Dutch national CRC screening in 2014 (the first year of introduction) was even higher, 68%. The investigators expect that 80% of these persons will fill out the familial risk questionnaire, resulting in 3.264 persons who perform both tests. As the investigators recommend invitees to perform the questionnaire in addition to FIT, the investigators assume that the percentage of persons only filling out the questionnaire and not performing FIT are negligible. Based on previous screening studies using a FIT positivity cut-off value of 50 ng Hb/mL for the OC-Sensor, it is assumed that 8% of these participants have a positive FIT result. In the current Dutch screening program, a different FIT is used (FOB-Gold) with a cut-off value of 275 ng Hb/ml. The FIT positivity rate with this test and with this cut-off value is unknown. However, a governmental announcement recently reported that the positivity rate is expected to remain 8% with this cut-off value. Therefore, the investigators expect 326 FIT positives in this study (8% of 4.080). Based on previous studies, approximately 40% of all persons with a positive FIT result will have advanced neoplasia. In our sample this concerns 130 persons. The percentage of persons with a familial CRC risk requiring surveillance colonoscopies in a screening population varies between 2.3% and 4%. Differences in the definition of an increased familial CRC risk could explain the variability in reported numbers. As the investigators are using a relatively large range in criteria for fulfilling the definition of a familial CRC risk, the highest reported percentage (4%) is assumed, which concerns 131 persons. The previously developed family history questionnaire has a sensitivity of 90% and 100% in identifying those persons qualifying for referral, in two subsequent validation phases respectively. For the purpose of this study, this validated questionnaire is adjusted to the recently renewed referral criteria. The investigators make the assumption that the questionnaire can identify all persons with a familial CRC syndrome based on referral criteria. Persons with a familial CRC syndrome who do not fulfill these criteria will be missed. This concerns an unknown number and will not be taken into account. A previous screening study showed that 6% of those with a positive FIT have an increased familial CRC risk. One can calculate that 3.8% of persons with a negative FIT have a familial CRC risk: 4% minus 6% of 8% (FIT positives), divided by 92% (FIT negatives). If one assumes that there is no difference in familial CRC risk between those who do and those who do not fill out the questionnaire, this involves 114 of 3.264 persons. Based on unpublished data by this research group it is estimated that 10% of those with a negative FIT have a familial CRC risk: 11 persons (10% of 114). A similar percentage was found in another screening study. Additionally, all participants with a familial CRC syndrome will be offered surveillance recommendations. In this sample, 131 persons are estimated to have a familial CRC syndrome. Of these, 16 persons (12%) will undergo a colonoscopy due to a positive FIT (6% of 8% FIT positives) and their familial CRC risk could be addressed at their visit to a colonoscopy center. The other 115 persons (88%) are expected to have a negative FIT and these persons (and their family members) would otherwise be unlikely to be identified as having a familial CRC syndrome.

ELIGIBILITY:
Inclusion Criteria: Six thousand persons eligible for the national CRC screening program, consisting of persons from the birth years 1941, 1945, 1953, 1955 and 1957 will be selected. These persons will be selected from four areas in North-Holland that are considered representative of the Netherlands regarding ethnical distribution and socioeconomic status: Aalsmeer, De Ronden Venen, Ouder-Amstel, Stichtse Vecht. These areas had an average participation-rate in 2014 that was comparable to the national participation rate (68.2%; a range from 65% to 75% is allowed). The distribution of age groups and gender will be comparable to the national screening distribution in 2016. Those who have been invited for a previous screening round in 2014 or for previous pilot-screening rounds will not be selected. In order to be eligible for participation, a subject must have been selected for participation in the national FIT-screening program in 2016.

Exclusion Criteria:

No specific exclusion criteria apply for participation in Family Matters, meaning that all invitees will receive a FIT as well as the questionnaire.

Ages: 59 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 1.5 years
  number of participants in whom advanced neoplasia is detected relative to the number of invitees

SECONDARY OUTCOMES:
Participation rate | 1.5 years
  Number of invitees completing the screening tests relative to the number of invitees
Positive predictive value | 1.5 years
  Number of participants in whom advanced neoplasia is detected, relative to the number of participants testing positive

OTHER OUTCOMES:
The number of invitees with a familial CRC syndrome | 1.5 years
FIT result of participants with a familial CRC syndrome | 1.5 years
The number of family members of participants with a familial CRC syndrome who receive an advice for genetic testing and/or surveillance colonoscopies | 1.5 years
The number of questionnaire participants who need help completing the questionnaire | 1.5 years
The number of persons with a positive questionnaire with a confirmed familial CRC syndrome | 1.5 years
The number of persons with a false-positive questionnaire as confirmed when verifying the completed questionnaire | 1.5 years
The number of persons with a false-negative questionnaire as confirmed when verifying the completed questionnaire in a random sample of those with a negative questionnaire | 1.5 years
Attendance rate to the intake visit at the department of clinical genetics | 1.5 years
Reasons for non-participation to genetic testing after a familial CRC risk | 1.5 years
  This will be analyzed in a telephone interview
Attendance rate to the pre-colonoscopy consultation after a positive FIT or a familial CRC syndrome | 1.5 years
Reasons for non-participation to colonoscopy after a positive FIT or a familial CRC syndrome | 1.5 years
  This will be analyzed in a telephone interview
The number of persons with non-advanced lesions (SSA/P, hyperplastic polyps, non-advanced adenomas) after a positive FIT or a familial CRC syndrome | 1.5 years
Comparison of diagnostic yield in detecting advanced neoplasia of FIT with the national CRC screening yield | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Dekker, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roos VH, Kallenberg FGJ, van der Vlugt M, Bongers EJC, Aalfs CM, Bossuyt PMM, Dekker E. Addition of an online, validated family history questionnaire to the Dutch FIT-based screening programme did not improve its diagnostic yield. Br J Cancer. 2020 Jun;122(12):1865-1871. doi: 10.1038/s41416-020-0832-8. Epub 2020 Apr 20. PMID 32307443